CLINICAL TRIAL: NCT04487834
Title: Effects of Simethicone and Vivatlac Baby in Infantile Colic
Brief Title: Effects of Vivatlac Baby on Crying Behavior of Colicky Babies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The President Stanisław Wojciechowski State University of Applied Sciences in Kalisz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Kalisz 2020-01
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Infantile Colic
MeSH Terms: conditions — Colic | interventions — Simethicone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simethicone Solution (Active Comparator): Treatment with simethicone (Espumisan®, 100 mg/ml, Berlin-Chemie / Menarini Polska Sp z o.o., Warsaw, Poland) for four weeks. Simethicone was administered 3-6 times per day with each treatment comprising 6 drops of the 100 mg/ml emulsion.
  Interventions: Drug: Simethicone Solution
- Vivatlac Baby (Experimental): Treatment with one stick pack of the multi-strain synbiotic (Vivatlac® Baby, Vivatrex GmbH, Rees, Germany) per day for four weeks. Each stick pack of Vivatlac® Baby contains a total of 10^9 colony forming units (CFU) with equal CFU amounts of the following probiotic bacteria: L. acidophilus LA-14, L. casei R0215; L. paracasei Lpc-3; L. plantarum Lp-115; L. rhamnosus GG, L. salivarius Ls-33, B. lactis Bl-04, B. bifidum R0071, B. longum R0175 and 1.43 g of the prebiotic fructooligosaccharides.
  Interventions: Dietary Supplement: Vivatlac Baby

INTERVENTIONS:
Drug: Simethicone Solution — Oral daily treatment for four weeks
  Other Names: Simethicone
  Arms: Simethicone Solution
Dietary Supplement: Vivatlac Baby — Oral daily treatment for four weeks
  Other Names: Multistrain Synbiotic
  Arms: Vivatlac Baby

SUMMARY:
Open trial with two parallel arms, assessing the effects of Simethicone and Vivatlac Baby in babies diagnosed for infantile colic.

DETAILED DESCRIPTION:
Babies aged 3 to 6 weeks will be diagnosed for infantile colic using the Wessel's criteria. Study design will be open label with two parallel arms (Simethicone and Vivatlac Baby). Vivatlac Baby is a synbiotic product containing probiotic bacteria (six lactobacilli and 3 bifidobacteria). Effects of treatments on crying behavior will be assessed by using parental 24h paper diaries.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed for infantile colic according to Wessel's criteria

Exclusion Criteria:

* previous treatment with probiotic or synbiotic
* previous treatment with antibiotics

Ages: 3 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Krauss, Prof., Principal Investigator — University of Applied Sciences in Kalisz, Poland
Locations (2):
- Poland (2):
  - GP Practice Pro Familia, Koziegłowy
  - Medical University in Poznań, Poznan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piatek J, Krauss H, Ciechelska-Rybarczyk A, Bernatek M, Wojtyla-Buciora P, Sommermeyer H. In-Vitro Growth Inhibition of Bacterial Pathogens by Probiotics and a Synbiotic: Product Composition Matters. Int J Environ Res Public Health. 2020 May 11;17(9):3332. doi: 10.3390/ijerph17093332. PMID 32403297
- [Derived] Piatek J, Bernatek M, Krauss H, Wojciechowska M, Checinska-Maciejewska Z, Kaczmarek P, Sommermeyer H. Effects of a nine-strain bacterial synbiotic compared to simethicone in colicky babies - an open-label randomised study. Benef Microbes. 2021 Jun 15;12(3):249-257. doi: 10.3920/BM2020.0160. Epub 2021 Mar 26. PMID 33765904
- See also: In-Vitro Growth Inhibition of Bacterial Pathogens by Probiotics and a Synbiotic: Product Composition Matters — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7246756/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 915 patients were assessed for eligibility.
Pre-assignment Details: 828 patients were excluded before randomization (parents of 704 patients declined to participate, 123 patients were diagnosed non-colic, 1 patient was excluded because of antibiotic treatment). 87 patients were randomized (33 to the Simethicone arm and 54 to the multi-strain synbiotic arm)
Groups:
- Multilac Baby: Treatment with one stick pack of the multi-strain synbiotic (Multilac® Baby, Vivatrex GmbH, Aachen, Germany) per day for four weeks. Each stick pack of Multilac® Baby contains a total of 10^9 colony forming units (CFU) with equal CFU amounts of the following probiotic bacteria: L. acidophilus LA-14, L. casei R0215; L. paracasei Lpc-3; L. plantarum Lp-115; L. rhamnosus GG, L. salivarius Ls-33, B. lactis Bl-04, B. bifidum R0071, B. longum R0175 and 1.43 g of the prebiotic fructooligosaccharides.
  Multilac Baby: Oral daily treatment for four weeks
Period: Overall Study
Arm/Group | Simethicone Solution | Multilac Baby
Started | 33 | 54
Completed | 33 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simethicone Solution | Vivatlac Baby | Total
Number analyzed (Participants) | 33 | 54 | 87
Age, Continuous [Mean (Standard Deviation); unit: days] — Age in days at enrollment
  days | 25.0 (1.9) | 26.0 (1.8) | 25.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 29 | 47
  Male | 15 | 25 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Poland | 33 | 54 | 87
Type of delivery [Count of Participants; unit: Participants] — (normal/caesarean)
  Participants
    Normal | 24 | 39 | 63
    Caesarean | 9 | 15 | 24
Birthweight [Mean (Standard Deviation); unit: g] — Birthweight in g
  g | 3480 (412) | 3500 (404) | 3492 (347)
Feeding [Count of Participants; unit: Participants] — breast/formula/mixed
  Participants
    Breast feeding | 22 | 27 | 49
    Formula feeding | 11 | 17 | 28
    Mixed feeding | 0 | 10 | 10
Days of crying [Mean (Standard Deviation); unit: days] — Days of crying last 3 weeks before start of treatment
  days | 18.2 (1.7) | 18.3 (2.1) | 18.2 (1.6)
Duration of evenning crying [Mean (Standard Deviation); unit: h/day] — Duration of evenning crying in three weeks before start of treatment
  h/day | 2.7 (0.5) | 2.8 (0.7) | 2.8 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction of Days Crying Equal or More Than 50 Percent From Baseline
Description: Measurement of days of crying during last three weeks before enrollment and before the end of treatment. Treatment success was determined by calculation the percentage of patients for whom the measurement was reduced by the respective treatment by equal or more than 50 percent, compared to the value at the time of enrollment.
Time Frame: Three weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Simethicone Solution | Vivatlac Baby
Number analyzed (Participants) | 33 | 54
Participants | 6 | 39
Statistical Analysis 1: Comparison: Simethicone Solution vs Vivatlac Baby; Test type: Superiority; p < 0.0001, Fisher Exact

2. Primary Outcome: Number of Participants With a Reduction of Average Duration of Evening Crying Equal or More Than 50 Percent
Description: Measurement of average duration of evening crying during last three weeks before enrollment and before the end of treatment. Treatment success was determined by calculation the percentage of patients for whom the measurement was reduced by the respective treatment by equal or more than 50 percent, compared to the value at the time of enrollment.
Time Frame: Three weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Simethicone Solution | Vivatlac Baby
Number analyzed (Participants) | 33 | 54
Participants | 13 | 46
Statistical Analysis 1: Comparison: Simethicone Solution vs Vivatlac Baby; Test type: Superiority; p = 0.0001, Fisher Exact

3. Primary Outcome: Number of Participants With a Reduction of Average Number of Crying Phases Per Day Equal or More Than 50 Percent
Description: Measurement average number of crying phases per day during last three weeks before enrollment and before the end of treatment. Treatment success was determined by calculation the percentage of patients for whom the measurement was reduced by the respective treatment by equal or more than 50 percent, compared to the value at the time of enrollment.
Time Frame: Three weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Simethicone Solution | Vivatlac Baby
Number analyzed (Participants) | 33 | 54
Participants | 14 | 27
Statistical Analysis 1: Comparison: Simethicone Solution vs Vivatlac Baby; Test type: Superiority; p = 0.4852, Fisher Exact

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Adverse events were collected by a non-systematic assessment: Every event considered by parents of babies to be an adverse event was reported as an event.
Arm/Group | Simethicone Solution | Multilac Baby
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/54
Other Adverse Events (participants affected / at risk) | 0/33 | 0/54

LIMITATIONS AND CAVEATS:
A limitation of the study is the use of parental diaries to measure infants' crying behavior. Using paper diaries is not without problems. Nevertheless, it has been shown that paper diary recordings of common infant behavior can provide reasonably good estimates of durations, while behavioral frequencies may be underestimated. Another major limitation of the study is that medication was not blinded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: Effects of Simethicone and Multilac Baby in Infantile Colic (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04487834/Prot_000.pdf
  • Study Protocol: Annex Patient Assessment Sheet Day 0 (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04487834/Prot_001.pdf
  • Study Protocol: Annex 24 Hours Parental Diary Form (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04487834/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04487834/SAP_003.pdf